CLINICAL TRIAL: NCT01861379
Title: The Role of Ghost Ileostomy in Laparoscopic Rectal Resection
Acronym: GILRR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Saverio Mari, Research Fellow, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DS-008
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Colo-rectal Anastomosis Dehiscence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ghost Ileostomy (Experimental): The patients were subjected to laparoscopic anterior rectal resection with performance of ghost ileostomy
  Interventions: Procedure: Ghost Ileostomy
- No protective stoma (Placebo Comparator): The patients were subjected to laparoscopic anterior rectal resection without simultaneous construction of any protective stoma.
  Interventions: Procedure: Ghost Ileostomy

INTERVENTIONS:
Procedure: Ghost Ileostomy — At the end of Laparoscopic Anterior Rectal Resection, once the colorectal anastomosis was performed, the terminal ileum was identified and a window in the mesentery was created to pass a rubber tube (we usually use an urinary catheter) around the intestinal loop. The tube was subsequently exteriorized trough the trocar incision in the right flank.
  Other Names: Virtual Ileostomy

SUMMARY:
To evaluate if the Ghost Ileostomy is really advantageous in laparoscopy we conducted a prospective randomized controlled study comparing 2 groups of patients undergoing anterior resection of the rectum laparoscopically. In the first group of patients at the end of the procedure was always performed a Ghost Ileostomy while in the second group no protective stoma was built at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Surgical Indication for Laparoscopic Anterior Rectal Resection
* Medium risk of anastomotic leakage

Exclusion Criteria:

* High risk of anastomotic leakage
* Lower risk of anastomotic leakage
* Advanced neoplasia (T4)
* Indication for inter-sphincteric resection hydro-pneumatic test of the anastomosis tightness showed positive for air leak
* Surgical procedure intraoperatively modified from the standard laparoscopic anterior rectal resection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2007-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Presence of Clinical Evident Anastomotic Leak | 15 days

SECONDARY OUTCOMES:
Postoperative complication | 15 days
Ghost Ileostomy complications | 15 days